CLINICAL TRIAL: NCT05662813
Title: a Phase II Studay to Assess the Efficacy and Safety of Almonertinib Therapy in Patients With Abnormal Liver Function After First/Second Generation TKI Treatment, or Almonertinib First-line Therapy in Patients With Basic Hepatopathy
Brief Title: Almonertinib Therapy in Patients With Abnormal Liver Function After EGFR-TKI Treatment, or Almonertinib First-line Therapy in Patients With Basic Hepatopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, LUO FENG, Study Chair, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022 Annual Review No.746
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR; NSCLC; abnormal liver function; hepatopathy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Liver Diseases; Digestive System Diseases | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Almonertinib (Experimental): Almonertinib 110 mg，orally once a day. Patients receive Almonertinib treatment until disease progression, unacceptable toxicity or other discontinuation criteria.
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib 110mg p.o qd. Patients receive Almonertinib treatment until disease progression, unacceptable toxicity or other discontinuation criteria.
  Other Names: HS-10296

SUMMARY:
To assess the efficacy and safety of Almonertinib therapy in patients with abnormal liver function after first/second generation EGFR-TKI treatment, or Almonertinib first-line therapy in patients with basic hepatopathy and locally advanced or metastatic EGFR-mutant non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a single arm, open-lable, phase II clinical trial，aimed to assess the efficacy and safety of Almonertinib therapy in EGFR-mutant advanced non-small cell lung cancer patients with abnormal liver function after the first/second generation EGFR-TKI treatment or EGFR-mutant advanced non-small cell lung cancer patients with basic hepatopathy and have not received any systematic treatment. The patients meet all the inclusion criterias, and do not meet any exclusion criteria can be included, the duration of patient observation is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* Locally advanced (IIIB and IIIC) or metastatic (IV) NSCLC.
* Tumor tissue samples or blood samples are confirmed to be EGFR sensitive mutations (including exon 19 deletion or L858R, both alone or coexist with other EGFR mutations).
* Patients have been treated with one kind of EGFR-TKIs and suffered from drug-induced liver injury, and have stopped EGFR-TKIs treatment before enrollment; or patients with basic hepatopathy (alcoholic liver disease, viral liver disease, metabolism related fatty liver disease, autoimmune liver disease, genetic metabolic liver disease), and patients can be treated with EGFR-TKIs after medical specialist evaluation, and no longger treated with hepatoprotective drugs (anti-inflammatory drugs, liver cell membrane repair protective agents, detoxification drugs, antioxidant drugs, cholagogic drugs) for 4 weeks before enrollment.
* ALT and AST ≤ 3 ULN, Child-Pugh grade A or B (≤ 9 points), and maintained for 4 weeks before enrollment (liver function evaluation criteria according to CTCAE 5.0) .
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3, and has not deteriorated at least 2 weeks, and the expected survival period is not less than 12 weeks.
* According to RECIST1.1, the patient has at least one intracranial target lesion and one extracranial target lesion. The requirements for target lesions are: measurable lesions that have not undergone local treatment such as irradiation or have clearly progressed after local treatment, with the longest diameter at baseline ≥10 mm (if it is a lymph node, the maximum short diameter is required to be ≥15 mm).

Exclusion Criteria:

* As judged by the investigator, patients with any serious or poorly controlled systemic diseases, such as poorly controlled hypertension, active bleeding-prone constitution, or active infection.
* Patients with any other malignant tumor in the past 5 years.
* Patients with prior drug-induced liver injury other than EGFR-TKIs.
* Patients with refractory nausea, vomiting or chronic gastrointestinal diseases, cannot swallow the study drug or who have received extensive intestinal resection, may affect the full absorption of Almonertinib.
* A history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of radiation pneumonitis requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
* Before Almonertinib treatment, patients with unresolved residual toxicity from previous anti-tumor therapy greater than CTCAE level 3, except for hair loss.
* Meet any of the following cardiac examination results:

  1. The average value of QT interval (QTcF) corrected by Fridericia's formula obtained from 3 ECG examinations at rest> 470 msec;
  2. Resting ECG suggests that there are various clinically significant rhythms, conduction or ECG morphological abnormalities that are judged by the investigator (such as complete left bundle branch block, 3 degree atrioventricular block, 2 degree atrium Ventricular block and PR interval> 250 msec, etc.);
  3. There are any factors that increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death or prolonged QT of immediate family members under 40 Any concomitant drugs in the interval;
  4. Left ventricular ejection fraction (LVEF) <50%.
* Insufficient bone marrow reserve or organ function, reaching any one of the following laboratory limits (no corrective treatment within 1 week before laboratory examination of blood draw):

  1. Absolute neutrophil count <1.5×109 / L;
  2. Platelet count <100×109 / L;
  3. Hemoglobin <90 g/L (<9 g/dL);
  4. Creatinine>1.5×ULN and creatinine clearance rate<50 mL/min (calculated by Cockcroft-Gault formula); Only when creatinine>1.5×ULN, creatinine clearance rate needs to be confirmed;
  5. Serum albumin (ALB) <28 g/L.
* Female with positive blood or urine pregnancy test results during lactation or within 3 days before the first administration of the study treatment.
* Active fungal, bacterial and/or viral infections requiring systemic treatment.
* Have a history of hypersensitivity to any active or inactive ingredients of Almonertinib or to drugs with similar chemical structure to Almonertinib or the same class of Almonertinib.
* Patients with decompensated cirrhosis, hepatic encephalopathy, hepatorenal syndrome, esophageal and gastric varices bleeding, and intractable ascites.
* Patients have treated with other three generations of EGFR-TKIs.
* Patients with any serious or uncontrolled disease, investigator judged that there are any patients with conditions that endanger the safety of the patient or interfere with the evaluation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months.
  ORR is defined as the number of patients with at least 1 visit response of CR (Complete response) or PR (Partial response) according to RECIST 1.1.

SECONDARY OUTCOMES:
Liver Safety | From the screening period to 28 days after treatment completion.
  Liver function indicators, including ALT, AST, TBIL, D-BIL, I-BIL, ALP, GGT, bile acid, ALB, GLB.
Progression-free survival | 24 months.
  PFS is defined as the time from date of enrollment until the date of disease progression as assessed according to RECIST 1.1 or death from any cause on study.
Disease control rate | 24 months.
  Disease control rate (DCR) is defined as the percentage of participants with disease control best overall response (complete response, partial response or stable disease).
Overall survival | From baseline until death due to any cause,up to a maximum of approximately 4 years.
  OS is defined as time from date of enrollment until date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Luo, Study Chair — West China Hospital; Yanyang Liu, Principal Investigator — West China Hospital; Zhixi Li, Principal Investigator — West China Hospital; Jiewie Liu, Principal Investigator — West China Hospital; Li Wang, Principal Investigator — West China Hospital; Jiantao Wang, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No